CLINICAL TRIAL: NCT05739188
Title: An Investigator-initiated Trial Evaluating the Efficacy and Safety of Anti-GPRC5D CAR-T Cells Therapy in the Treatment of Relapsed / Refractory(r/r) Multiple Myeloma(MM)
Brief Title: Safety and Efficacy of Anti-GPRC5D CAR-T Cells Therapy in the Treatment of r/r MM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-22-012
Record Dates: First submitted 2023-02-04; First posted 2023-02-22 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: CAR-T; GPRC5D
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This is a"3+3"dose escalation study, in which three dose groups are set three different dose levels of CAR-T cells:
  Dose level one: 3.0×10^6 /kg±20%; Dose level two:6.0×10^6 /kg±20%; Dose level three:1.0×10^7 /kg±20%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-GPRC5D CAR-T (Experimental): Subjects who meet the enrollment conditions will receive intravenous infusion of anti--GPRC5D CAR-T Cells after lymphodepleting therapy.
  Interventions: Biological: Anti-GPRC5D CAR-T cells infusion

INTERVENTIONS:
Biological: Anti-GPRC5D CAR-T cells infusion — This is a"3+3"dose escalation study, in which three dose groups are set three different dose levels of CAR-T cells:
  Dose level one: 3.0×10^6 /kg±20%; Dose level two:6.0×10^6 /kg±20%; Dose level three:1.0×10^7 /kg±20%.

SUMMARY:
It is a single-center, open-labeled, single-arm, non-randomized investigator-initiated trial evaluating the efficacy and safety of anti-GPRC5D CAR-T cells therapy for relapsed and refractory(r/r) multiple myeloma(MM).

DETAILED DESCRIPTION:
This open label, single-arm, Phase I study aims to evaluate the efficacy and safety of Anti-GPRC5D CAR-T in subjects with relapsed and refractory(r/r) multiple myeloma(MM). A leukapheresis procedure will be performed to manufacture Anti-GPRC5D chimeric antigen receptor (CAR) modified T cells. Prior to Anti-GPRC5D CAR-T cells infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide. After infusion, the safety and efficacy of CAR-T therapy was evaluated by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian understands and voluntarily signs the informed consent, and is expected to complete the follow-up examination and treatment of the study procedure;
2. Age 18-75 years old, gender unlimited;
3. Patients diagnosed with multiple myeloma according to International Myeloma Working Group(IMWG) diagnostic criteria;
4. Subjects who had failed treatment with at least 3 drugs of different mechanisms (including chemotherapy, proteasome inhibitors, immunomodulators, etc.), or had progressed or relapsed during the last treatment period or within 6 months after the end of treatment;
5. The presence of measurable lesions at screening was determined according to any of the following criteria, defined as: (1) serum monoclonal immunoglobulin (M-protein) level ≥1.0 g/dL; (2) urine M protein level ≥200 mg/ 24h; (3) Light chain multiple myeloma diagnosed with no measurable lesion in serum or urine: serum immunoglobulin free light chain ≥10 mg/dL and serum immunoglobulin κ/γ free light chain ratio abnormal;
6. The patient has recovered from the toxicity of the prior treatment, i.e., CTCAE toxicity grade < 2 (unless the abnormality is related to the tumor or is stable as judged by the investigator and has little impact on safety or efficacy);
7. Eastern cooperative oncology group (ECOG) score is 0-2;
8. Survival is expected to be greater than 3 months;
9. Adequate liver , kidney and cardiopulmonary function;
10. Willingness to complete the informed consent process and to comply with study procedures and visit schedule.

Exclusion Criteria:

1. Have been diagnosed with or treated for aggressive malignancies other than multiple myeloma;
2. Prior antitumor therapy (prior to blood collection for CAR-T preparation) : targeted therapy, epigenetic therapy, or investigational drug therapy within 14 days or at least 5 half-lives, whichever is shorter;
3. It is suspected that MM has involved the central nervous system or meninges and has been confirmed by MRI or CT, or there are other active central nervous system diseases;
4. Clinically significant central nervous system diseases, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, psychosis, active central nervous system involvement or cancerous meningitis;
5. HBsAg or HBcAb are positive, and the quantitative detection of hepatitis B virus(HBV) DNA in peripheral blood is more than 100 copies / L;hepatitis C virus (HCV) antibody and HCV RNA in peripheral blood are positive; HIV antibody positive; Syphilis antibody is positive in the first screening;
6. Pregnant or breastfeeding;
7. Severe active viral, bacterial or uncontrolled systemic fungal infections; Hereditary bleeding / coagulation diseases, history of non traumatic bleeding or thromboembolism, other diseases that may increase the risk of bleeding, etc;Patients who received autologous hematopoietic stem cell transplantation (ASCT) within 8 weeks before screening, or who plan to undergo ASCT during the study period;
8. Any unstable systemic disease: including but not limited to unstable angina, cerebrovascular accident or transient cerebral ischemia (within 6 months before screening), myocardial infarction (within 6 months before screening), congestive heart failure [New York Heart Association (NYHA) classification ≥ grade III], severe arrhythmia with poor drug control, liver, kidney or metabolic diseases;
9. Had hypersensitivity or intolerance to any drug used in this study;
10. Persons with serious mental illness;
11. Alcoholics or persons with a history of drug abuse;
12. Systemic diseases judged by researchers to be unstable: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
13. Patients with acute/chronic graft-versus-host disease (GVHD) or requiring immunosuppressive therapy for GVHD within 6 months prior to screening;
14. Any unsuitable to participate in this trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Up to 12 months after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included. Description, time, classification, and outcome of AE events resulted from the investigational medical product, delivery method, or emergency measures will be recorded in the case report form.
Dose limited toxicity (DLT) | Up to 1 month after infusion
  Dose limited toxicity(DLT) was defined as the occurrence of any of the following adverse events within 28 days of the infusion of CAR-T cells after optimal supportive treatment, which were discussed with the investigator and determined to be associated or likely to be associated with the infusion.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years after infusion
  Overall Response Rate (ORR) is defined as the proportion of subjects achieving strict complete remission(sCR), complete response(CR), very good partial response(VGPR） and partial response(PR).
Concentration of CAR-T cells | Days 4, 7, 10, 14 and months 2, 3, 6, 9, 12 after infusion
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion
Progression-free survival(PFS) | Up to 2 years
  Progression-free survival(PFS) refers to the time from cell reinfusion to the first assessment of tumor progression or death from any cause.
Overall survival(OS) | Up to 2 years
  Overall survival (OS) refers to the time from the time the patient received an infusion of CAR-T cells until death (from any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (2):
- China (2):
  - 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan
  - No.212 Daguan Road, Xishan District, Kunming, Yunnan